CLINICAL TRIAL: NCT01089673
Title: A Retrospective Study of the Effects of Molecular Diagnostics on Wound Care Outcomes
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-016
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Wounds
Keywords: retrospective data collection
MeSH Terms: conditions — Wounds and Injuries | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: retrospective data analysis
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — retrospective data collection

SUMMARY:
A retrospective molecular diagnostic review on wound care outcomes between two time periods. The time periods include June, July, August of 2008 and June, July, August of 2009. The retrospective review would analyze the days of healing during those two timeframes, upon the introduction of molecular diagnostic testing.

ELIGIBILITY:
Inclusion Criteria:

* A patient record captured during June, July, August 2008 and June, July, or August of 2009.

Exclusion Criteria:

* A patient record captured outside the time frame of June, July August 2008 or June, July, August of 2009.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient records would be extracted from the electronic health record system of Southwest Regional Wound Care Center.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
A retrospective molecular diagnostic review on wound care outcomes between two time periods. | The time periods include June, July, August of 2008 and June, July, August of 2009.
  The retrospective review would analyze the days of healing during those two timeframes, upon the introduction of molecular diagnostic testing.